CLINICAL TRIAL: NCT01791686
Title: A Pilot, Open-label, Multicenter Clinical Trial of CDX-1135 in Pediatric and Adult Patients With Dense Deposit Disease
Brief Title: Clinical Trial of CDX-1135 in Pediatric and Adult Patients With Dense Deposit Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio prioritization due to slow enrollment and variable spectrum of potential complement abnormalities in DDD patients.
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1135-01
Record Dates: First submitted 2013-01-29; First posted 2013-02-15 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Dense Deposit Disease; Membranoproliferative Glomerulonephritis Type II; C3 Glomerulonephritis
Keywords: Dense Deposit Disease; DDD
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dense Deposit Disease (Experimental): ► Induction Period
  Patients will receive CDX-1135 as an IV infusion twice weekly (Mon-Thur or Tues-Fri). There will be two doses of 5 mg/kg, with intrapatient dose-escalation in 5 mg/kg increments up to a maximum dose of 30 mg/kg. This period may last up to 8 weeks.
  ► Maintenance Period
  The starting dose for CDX-1135 Maintenance will be the same dose level as the last dose during the Induction Period; however, the Maintenance Period allows for dose decrease to 2 mg/kg, which is lower than the starting dose in the Induction Period.
  Patients will receive CDX-1135 as an IV infusion twice weekly (Mon-Thur or Tues-Fri) for up to a total of 26 weeks.
  Interventions: Drug: CDX-1135

INTERVENTIONS:
Drug: CDX-1135
  Other Names: TP10; sCR1

SUMMARY:
This study is evaluating the study drug (CDX-1135) in patients with dense deposit disease (DDD). The objective is to evaluate the safety and activity of repeated doses of CDX-1135 in pediatric and adult patients with DDD. After screening, eligible patients will be entered into the Induction Period. The Induction Period is up to 4 weeks. Following normalization of complement activity, patients will enter into the Maintenance Period.The total treatment duration is up to 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must be

1. Patient and/or parent/legal guardian (as appropriate) must give written informed consent
2. Four (4) years of age or older
3. Must have DDD, confirmed by renal biopsy within 6 months of study enrollment (Confirmation by University of Iowa investigators is required). If the patient is post transplant, the repeat renal transplant biopsy must show C3 dominant glomerulonephritis, and the patient must have a history of known DDD in the native kidney
4. Signs of abnormal complement pathway activity
5. Serum creatinine level must be abnormal
6. Screening lab values criteria:

   1. Hgb ≥ 9.0 g/dL
   2. Platelets ≥ 100,000/mm^3
   3. ALT and AST ≤ 3.0 x upper limit of normal
   4. C3 serum <50% of the lower limit of normal
   5. 24 hour urine protein >1000 mg/day, or urine protein:creatinine ratio >1.0
7. Both male and female patients of childbearing potential enrolled must use adequate birth control during the trial and for 1 month after stopping study drug
8. Willing and able to comply with study procedures, including pre-study vaccinations (meningitis, haemophilus and pneumococci) and agree to a renal biopsy at Week 13 and at the end of the study
9. Any anti-proteinuric medications (eg, angiotensin converting enzyme inhibitors, angiotensin II receptor blockers) must be at a stable dose for 4 weeks prior to first dose of CDX-1135

Exclusion Criteria:

Among other criteria, patients must not be

1. Dialysis or a low estimated glomerular filtration rate <30 ml/min/1.73m^2 over a 4-week period prior to Screening
2. Active or untreated systemic bacterial infection
3. Pregnant or lactating
4. Rituximab therapy (unless discontinued with B cell levels and immunoglobulin levels normalized by study entry)
5. Immunosuppressive therapies (except for low dose steroids [≤10 mg per day] given for non-DDD related conditions such as asthma). Exceptions will be made for renal transplant patients, who may receive any appropriate therapies as needed to maintain the transplant (i.e., to prevent rejection)
6. Treatment with any complement inhibitor within 3 months of study entry or any other investigational drug, device, or experimental procedure within 4 weeks prior to enrollment
7. For renal transplant patients only: histology findings of treatable rejection (i.e. that the usual transplant physician would seek to treat). Chronic allograft nephropathy is not exclusionary provided the patient's glomerular filtration rate meets other entry criteria
8. Preexisting condition with an association as a potential cause of DDD (i.e., Monoclonal Gammopathy of Undetermined Significance) or an alternate glomerular disease
9. Cancer except for adequately treated and cured basal or squamous cell skin cancer, curatively treated in situ disease, or other cancer that the patient has been disease-free for ≥ 5 years
10. Myocardial infarction within 1 year of screening, congestive heart failure, arrhythmia persistent on medication at screening or chronic lung disease
11. Known HIV, Hepatitis B or Hepatitis C
12. Any medical or psychological condition that would increase the patient's risk by being in this study or would interfere with interpretation of the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety | From first study drug dose for up to 26 weeks
  * Incidence and severity of adverse events (AE) will be assessed at every visit. AEs and serious adverse events (SAEs) will be assessed from the first dose of study drug through 33 days after the last dose
  * To evaluate the safety of repeated dosing in patients with DDD. Safety will be assessed based on changes in clinical laboratory tests, physical exams, vital signs, ophthalmic exams and ECGs [for patients ≥ 35 years of age].
C3 and AP Normalization | Regular assessments from study start up to 26 weeks
  The proportion of patients with normalization of serum C3, serum C3 breakdown products, or alternative pathway (AP) complement activity. These blood tests will be assessed on each dosing day and upon Study Completion /Termination.

SECONDARY OUTCOMES:
Duration of and time to normalize C3 and AP | Regular assessments from study start up to 26 weeks
  Time to normalization of serum levels of C3 or C3 breakdown products and duration of normalization and assays of alternative pathway activity. These blood tests will be assessed on each dosing day and upon Study Completion /Termination.
Renal Function | Regularly from study start up to 26 weeks
  Stabilization and/or improvement in renal function (as measured by serum creatinine and proteinuria). These lab tests will be performed weekly during the Induction Period, monthly during the Maintenance Period and upon Study Completion /Termination.
Renal biopsy | Occurs up to 3 times from study start up to 26 weeks
  Improvement on renal biopsy (as measured by reduction in C3 deposition in the glomerular basement membrane). This biopsy may be performed during screening, week 13, and upon Study Completion /Termination.
Immunogenicity | Regular assessments from study start up to 26 weeks
  Immunogenicity (development of antibodies to CDX-1135). This sample will be collected prior to dosing on Week 1, monthly during treatment, and upon Study Completion /Termination

OTHER OUTCOMES:
CDX-1135 concentrations | Regular assessments from study start up to 26 weeks
  Serum concentrations of CDX-1135 will be determined from blood samples collected prior to dosing and post-dosing. (on each dosing day)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Nester, MD, MSA, Principal Investigator — University of Iowa; Richard Smith, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States